CLINICAL TRIAL: NCT05299060
Title: Effectiveness of Cyanoacrylate Glue in the Fixation of Midline and Peripherally Inserted Central Catheters in Hospitalized Adult Patients: Randomised Clinical Trial (CIANO-ETI)
Acronym: CIANO-ETI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Arnau de Vilanova (Other)
Responsible Party: Principal Investigator, Ferran Padilla Nula, Principal Investigator, Hospital Arnau de Vilanova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01-20
Record Dates: First submitted 2022-02-26; First posted 2022-03-28 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Vascular Access Device; Catheterization, Peripheral; Nursing Care; Randomized Controlled Trial
Keywords: Cyanoacrylates; Cyanoacrylate; Tissue adhesive

STUDY DESIGN:
Intervention Model Description: Classical parallel model with an intervention group, to which cyanoacrylate tissue adhesive was applied, and a control group.
Who Masked: Participant, Care Provider
Masking Description: The investigators are the ones who performed the insertion of the catheters and the subsequent data collection, but neither the patients nor the healthcare staff knew which patient was wearing tissue adhesive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): After cannulation of a midline catheter or peripherally inserted central venous catheter with modified micro-Seldinger technique, the control group underwent standard care.
  Interventions: Procedure: standard cure
- Intervention (Experimental): After cannulation of a midline catheter or peripherally inserted central venous catheter with a modified micro-Seldinger technique, the intervention group underwent the standard treatment plus application of cyanoacrylate tissue adhesive (SecurePortIV®) at the puncture site.
  Interventions: Procedure: cyanoacrylate adhesive (SecurePortIV®)

INTERVENTIONS:
Procedure: cyanoacrylate adhesive (SecurePortIV®) — Application of cyanoacrylate tissue adhesive (SecurePortIV®) to the puncture site plus standard wound care.
  Arms: Intervention
Procedure: standard cure — The standard cure consists of:
  * Application of hemostasis at the point of insertion for 2 minutes post puncture or until bleeding stops.
  * Fix with clear polyurethane dressing (3M®-1655 Tegaderm™ IV) and sutureless fixation device (BD-19940 StatLock™ PICC Plus).
  Arms: Control

SUMMARY:
Introduction: Venous access is increasingly necessary and essential in healthcare institutions, where more than 75% of hospitalised patients have some type of vascular access device cannulated. Due to their pathophysiological characteristics and pharmacological needs, some patients require special catheters, such as midline or peripherally inserted central catheters. In an attempt to reduce the main complications related to these, the safety of cyanoacrylate tissue adhesive has recently been demonstrated in the post-insertion treatment of vascular access devices.

Objective: To evaluate the efficacy of the use of cyanoacrylate tissue adhesive as fixation in the post-insertion of cannulated middle and central venous catheters with modified micro-Seldinger technique in acute hospitalized patients.

Methods: Randomised clinical trial with two groups(1:1): control and intervention. The control group received a cure with sutureless device plus transparent membrane and the intervention group received the same cure plus the cyanoacrylate glue. The study was approved by the Drug Research Ethics Committee of the Lleida health region. health region.

KEYWORDS: Cyanoacrylates; Vascular Access Device; Catheterization, Peripheral; Nursing Care; Randomized Controlled Trial.

DETAILED DESCRIPTION:
A randomized clinical study with two arms (control group and intervention group) was performed.

Patients were selected according to whether they met the inclusion/exclusion criteria and all patients who met the criteria were offered to participate on a voluntary basis. These were collected by the intravenous therapy team (ETI) of the Arnau de Vilanova University Hospital (HUAV) in Lleida, from September 16, 2020 until the completion of the collection of the total number of patients required for the study (n=216).

Patients required insertion of a midline venous catheter (BD-18580 PowerMidline™ 4F) or a peripherally inserted central catheter (BD-20178 PowerPICC™ 4,5 or 6 F), according to the ETI-HUAV algorithm. All insertions were performed with the aid of ultrasound as a guiding technique. In addition, all patients underwent dermatotomy during the technique and the application of a post-insertion hemostasis protocol for at least 2 minutes or until the insertion site stopped bleeding, in order to unify the researchers' criteria.

After insertion of the vascular access device, the control group underwent the standard dressing: transparent polyurethane dressing with reinforced edge (3M®-1655 Tegaderm™ IV) and Sutureless Fixation Device (BD-19940 StatLock™ PICC Plus); and the intervention group, the standard dressing plus application of cyanoacrylate tissue adhesive (SP-015V SecurePortIV™ from Adhezion Biomedical, Llc.).

Afterwards, 3 scheduled cures were performed, at 24 hours, 72 hours and 7 days post-insertion, looking for the main complications: bleeding and/or pericatheter exudate, catheter displacement, signs of phlebitis and catheter-related pain.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* requiring cannulation of a midline catheter (BD-18580 PowerMidline™ 4F) or a PICC (BD-20178 PowerPICC™ 4.5 or 6 F)
* who accepted and signed the informed consent voluntarily
* with an inpatient unit admission of minimum 7 days

Exclusion Criteria:

* patients with skin conditions contraindicating the application of a skin glue or known allergy to cyanoacrylate, as recorded in the clinical history

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | 7 days
  Percentage of participants with adverse events after being treated with cyanoacrylate tissue adhesive at the puncture site after insertion of cannulated middle and central venous catheters with the modified micro-Seldinger technique.

SECONDARY OUTCOMES:
Number of participants with post-treatment hemorrhage assessed by observation (yes/no). | 7 days
  Percentage of participants with pericatheter bleeding after puncture of a midline or central venous catheter with the modified micro-Seldinger technique. Four cures will be performed: post puncture, at 24 hours, 72 hours and 7 days, where the puncture site will be visualized for signs of bleeding and it will be noted whether there is bleeding or not.
Number of participants with post-treatment catheter displacement assessed by observation (yes/no). | 7 days
  Percentage of participants with catheter displacement after puncture of a midline or central venous catheter with the modified micro-Seldinger technique. Four cures will be performed: post puncture, at 24 hours, 72 hours and 7 days, where the puncture site will be visualized to check if the catheter is still in the same point or if it has been displaced.
Number of participants with post-treatment phlebitis assessed with the Maddox visual phlebitis rating scale. | 7 days
  Percentage of participants with phlebitis after puncture of a midline or central venous catheter with the modified micro-Seldinger technique. Four cures will be performed: post puncture, at 24 hours, 72 hours and 7 days, where the puncture site will be visualized to check for signs of phlebitis, according to the Maddox scale.
Number of participants with post-treatment pain in extremity assessed with the EVA scale. | 7 days
  Percentage of participants with pain in extremity after puncture of a midline or central venous catheter with the modified micro-Seldinger technique. Four cures will be performed: post puncture, at 24 hours, 72 hours and 7 days, where the patient will be asked what pain he/she feels in the extremity related to the catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Padilla-Nula, Principal Investigator — Arnau de Vilanova hospital
Locations (1):
- Hospital Universitari Arnau de Vilanova, Lleida, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Contact the principal investigator by mail: FPADILLA@gencat.cat
Supporting Information: Study Protocol
Time Frame: The data is already available, there is no time limit.
Access Criteria: Be a researcher or group of researchers.

REFERENCES:
- [Background] Alexandrou E, Ray-Barruel G, Carr PJ, Frost S, Inwood S, Higgins N, Lin F, Alberto L, Mermel L, Rickard CM. International prevalence of the use of peripheral intravenous catheters. J Hosp Med. 2015 Aug;10(8):530-3. doi: 10.1002/jhm.2389. Epub 2015 Jun 3. PMID 26041384
- [Background] Fabiani A, Eletto V, Dreas L, Beltrame D, Sanson G. Midline or long peripheral catheters in difficult venous access conditions? A comparative study in patients with acute cardiovascular diseases. Am J Infect Control. 2020 Oct;48(10):1158-1165. doi: 10.1016/j.ajic.2019.12.025. Epub 2020 Jan 21. PMID 31973988
- [Background] Kang J, Chen W, Sun W, Ge R, Li H, Ma E, Su Q, Cheng F, Hong J, Zhang Y, Lei C, Wang X, Jin A, Liu W. Peripherally inserted central catheter-related complications in cancer patients: a prospective study of over 50,000 catheter days. J Vasc Access. 2017 Mar 21;18(2):153-157. doi: 10.5301/jva.5000670. Epub 2017 Feb 8. PMID 28218366
- [Background] Bodenham A. Vascular acces. Rev Med Clin Condes [Internet]. 2017;28(5):701-12. Available from: http://dx.doi.org/10.1016/j.rmclc.2017.07.011
- [Background] Corley A, Marsh N, Ullman AJ, Rickard CM. Tissue adhesive for vascular access devices: who, what, where and when? Br J Nurs. 2017 Oct 26;26(19):S4-S17. doi: 10.12968/bjon.2017.26.19.S4. PMID 29068728
- [Background] Lacostena-Perez ME, Buesa-Escar AM, Gil-Alos AM. Complications related to the insertion and maintenance of peripheral venous access central venous catheter. Enferm Intensiva (Engl Ed). 2019 Jul-Sep;30(3):116-126. doi: 10.1016/j.enfi.2018.05.002. Epub 2018 Sep 3. English, Spanish. PMID 30190250
- [Background] Fujioka G, Newcomb P, Hunchusky C, Myers H, Behan D. Pain Perception of a Structured Vascular Access Team Approach to Short Peripheral Catheter (SPC) Placement Compared to SPC Placement by Bedside Nurses. J Infus Nurs. 2020 Jan/Feb;43(1):33-38. doi: 10.1097/NAN.0000000000000352. PMID 31876772
- [Background] Braga LM, Parreira PM, Oliveira ASS, Monico LDSM, Arreguy-Sena C, Henriques MA. Phlebitis and infiltration: vascular trauma associated with the peripheral venous catheter. Rev Lat Am Enfermagem. 2018;26:e3002. doi: 10.1590/1518-8345.2377.3002. Epub 2018 May 17. PMID 29791668
- [Background] Ellis ML, Okano S, McCann A, McDowall A, Van Kuilenburg R, McCarthy AL, Joubert W, Harper J, Jones M, Mollee P. Catheter-related thrombosis incidence and risk factors in adult cancer patients with central venous access devices. Intern Med J. 2020 Dec;50(12):1475-1482. doi: 10.1111/imj.14780. PMID 32043739
- [Background] Moureau N. Impact and Safety Associated with Accidental Dislodgement of Vascular Access Devices: A Survey of Professions, Settings, and Devices. JAVA - J Assoc Vasc Access. 2018 Dec 1;23(4):203-15.
- [Background] Nicholson J, Hill J. Cyanoacrylate tissue adhesive: a new tool for the vascular access toolbox. Br J Nurs. 2019 Oct 24;28(19):S22-S28. doi: 10.12968/bjon.2019.28.19.S22. PMID 31647725
- [Background] Chaves F, Garnacho-Montero J, Del Pozo JL, Bouza E, Capdevila JA, de Cueto M, Dominguez MA, Esteban J, Fernandez-Hidalgo N, Fernandez Sampedro M, Fortun J, Guembe M, Lorente L, Pano JR, Ramirez P, Salavert M, Sanchez M, Valles J. Diagnosis and treatment of catheter-related bloodstream infection: Clinical guidelines of the Spanish Society of Infectious Diseases and Clinical Microbiology and (SEIMC) and the Spanish Society of Spanish Society of Intensive and Critical Care Medicine and Coronary Units (SEMICYUC). Med Intensiva (Engl Ed). 2018 Jan-Feb;42(1):5-36. doi: 10.1016/j.medin.2017.09.012. English, Spanish. PMID 29406956
- [Background] Mihala G, Ray-Barruel G, Chopra V, Webster J, Wallis M, Marsh N, McGrail M, Rickard CM. Phlebitis Signs and Symptoms With Peripheral Intravenous Catheters: Incidence and Correlation Study. J Infus Nurs. 2018 Jul/Aug;41(4):260-263. doi: 10.1097/NAN.0000000000000288. PMID 29958263
- [Background] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee (HICPAC). Guidelines for the prevention of intravascular catheter-related infections. Clin Infect Dis. 2011 May;52(9):e162-93. doi: 10.1093/cid/cir257. Epub 2011 Apr 1. No abstract available. PMID 21460264
- [Background] Song IK, Kim EH, Lee JH, Jang YE, Kim HS, Kim JT. Seldinger vs modified Seldinger techniques for ultrasound-guided central venous catheterisation in neonates: a randomised controlled trial. Br J Anaesth. 2018 Dec;121(6):1332-1337. doi: 10.1016/j.bja.2018.08.008. Epub 2018 Sep 7. PMID 30442261
- [Background] Gorski LA, Hadaway L, Hagle ME, Broadhurst D, Clare S, Kleidon T, Meyer BM, Nickel B, Rowley S, Sharpe E, Alexander M. Infusion Therapy Standards of Practice, 8th Edition. J Infus Nurs. 2021 Jan-Feb 01;44(1S Suppl 1):S1-S224. doi: 10.1097/NAN.0000000000000396. No abstract available. PMID 33394637
- [Background] Simonova G, Rickard CM, Dunster KR, Smyth DJ, McMillan D, Fraser JF. Cyanoacrylate tissue adhesives - effective securement technique for intravascular catheters: in vitro testing of safety and feasibility. Anaesth Intensive Care. 2012 May;40(3):460-6. doi: 10.1177/0310057X1204000311. PMID 22577911
- [Background] Bugden S, Shean K, Scott M, Mihala G, Clark S, Johnstone C, Fraser JF, Rickard CM. Skin Glue Reduces the Failure Rate of Emergency Department-Inserted Peripheral Intravenous Catheters: A Randomized Controlled Trial. Ann Emerg Med. 2016 Aug;68(2):196-201. doi: 10.1016/j.annemergmed.2015.11.026. Epub 2015 Dec 31. PMID 26747220
- [Background] Rickard CM, Edwards M, Spooner AJ, Mihala G, Marsh N, Best J, Wendt T, Rapchuk I, Gabriel S, Thomson B, Corley A, Fraser JF. A 4-arm randomized controlled pilot trial of innovative solutions for jugular central venous access device securement in 221 cardiac surgical patients. J Crit Care. 2016 Dec;36:35-42. doi: 10.1016/j.jcrc.2016.06.006. Epub 2016 Jun 21. PMID 27546745
- [Background] Reynolds H, Taraporewalla K, Tower M, Mihala G, Tuffaha HW, Fraser JF, Rickard CM. Novel technologies can provide effective dressing and securement for peripheral arterial catheters: A pilot randomised controlled trial in the operating theatre and the intensive care unit. Aust Crit Care. 2015 Aug;28(3):140-8. doi: 10.1016/j.aucc.2014.12.001. Epub 2015 Jan 9. PMID 25583412
- [Background] Rickard CM, Marsh N, Webster J, Runnegar N, Larsen E, McGrail MR, Fullerton F, Bettington E, Whitty JA, Choudhury MA, Tuffaha H, Corley A, McMillan DJ, Fraser JF, Marshall AP, Playford EG. Dressings and securements for the prevention of peripheral intravenous catheter failure in adults (SAVE): a pragmatic, randomised controlled, superiority trial. Lancet. 2018 Aug 4;392(10145):419-430. doi: 10.1016/S0140-6736(18)31380-1. Epub 2018 Jul 26. PMID 30057103
- [Background] Biasucci DG, Pittiruti M, Taddei A, Picconi E, Pizza A, Celentano D, Piastra M, Scoppettuolo G, Conti G. Targeting zero catheter-related bloodstream infections in pediatric intensive care unit: a retrospective matched case-control study. J Vasc Access. 2018 Mar;19(2):119-124. doi: 10.5301/jva.5000797. Epub 2018 Feb 19. PMID 29148002
- [Background] Zhang S, Guido AR, Jones RG, Curry BJ, Burke AS, Blaisdell ME. Experimental study on the hemostatic effect of cyanoacrylate intended for catheter securement. J Vasc Access. 2019 Jan;20(1):79-86. doi: 10.1177/1129729818779702. Epub 2018 Jun 20. PMID 29923442
- [Background] Di Puccio F, Giacomarro D, Mattei L, Pittiruti M, Scoppettuolo G. Experimental study on the chemico-physical interaction between a two-component cyanoacrylate glue and the material of PICCs. J Vasc Access. 2018 Jan;19(1):58-62. doi: 10.5301/jva.5000816. PMID 29148010
- [Background] Maddox RR, Rush DR, Rapp RP, Foster TS, Mazella V, McKean HE. Double-blind study to investigate methods to prevent cephalothin-induced phlebitis. Am J Hosp Pharm. 1977 Jan;34(1):29-34. PMID 831472
- [Background] Huskisson EC, Jones J, Scott PJ. Application of visual-analogue scales to the measurement of functional capacity. Rheumatol Rehabil. 1976 Aug;15(3):185-7. doi: 10.1093/rheumatology/15.3.185. PMID 968347
- [Background] Babaieasl F, Yarandi HN, Saeidzadeh S, Kheradmand M. Comparison of EMLA and Diclofenac on Reduction of Pain and Phlebitis Caused by Peripheral IV Catheter: A Randomized-Controlled Trial Study. Home Healthc Now. 2019 Jan/Feb;37(1):17-22. doi: 10.1097/NHH.0000000000000704. PMID 30608463
- [Background] Goossens GA, De Waele Y, Jerome M, Fieuws S, Janssens C, Stas M, Moons P. Diagnostic accuracy of the Catheter Injection and Aspiration (CINAS) classification for assessing the function of totally implantable venous access devices. Support Care Cancer. 2016 Feb;24(2):755-761. doi: 10.1007/s00520-015-2839-x. Epub 2015 Jul 26. PMID 26209949